CLINICAL TRIAL: NCT02901704
Title: A Prospective, Multi-centers, Randomized,Controlled, Blinded,Superiority Trial of Renal Denervation Using Iberis MultiElectrode Renal Denervation System for the Treatment of Primary Hypertension.
Brief Title: Renal Denervation by Iberis MultiElectrode Renal Denervation System in Patients With Primary Hypertension
Acronym: Iberis-HTN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai AngioCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT201601
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- renal denervation (Experimental): Iberis Multielectrode Renal Denervation System (AngioCare)
  Interventions: Device: Renal Denervation System (AngioCare)
- Sham procedure (Sham Comparator): Renal anigography
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Device: Renal Denervation System (AngioCare) — After a renal angiography according to standard procedures, subjects remain blinded and are immediately treated with the renal denervation procedure after randomization.
  Arms: renal denervation
Procedure: Sham procedure — After a renal angiography according to standard procedures, subjects remain blinded and remain on the catheterization lab table for at least 10 minutes prior to introducer sheath removal.
  Arms: Sham procedure

SUMMARY:
The purpose of Iberis-HTN trial is to evaluate the safety and effectiveness of renal denervation in subjects with primary hypertension by using Iberis multielectrode renal denervation system

DETAILED DESCRIPTION:
The purpose was to evaluate 3-month outcomes of RDN for the treatment of primary hypertension in Chinese patients.In a prospective, multi-center study, 216 Chinese patients with primary hypertension would be recruited to undergo RDN by Iberis Multielectrode denervation system. The primary effectiveness endpoint wasReduction in average 24-hour ambulatory systolic blood pressue at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Primary Hypertension
* Stable medication regimen including 3 antihypertensive medications of different classes, including a diuretic (with no changes for a minimum of 4 weeks prior to screening) and 1) Office SBP ≥150 and ≤180 mmHg, and DBP ≥90 , 2) average 24-hour ambulatory systolic blood pressue and/or DBP ≥135 and ≤170 mmHg
* Main renal arteries with ≥3 mm diameter or with ≥20 mm treatable length (by visual estimation)
* Written informed consent

Exclusion Criteria:

Clinical Exclusion Criteria:

* Known secondary hypertension
* Type 1 diabetes mellitus
* Has an implantable cardioverter defibrillator (ICD) or pacemaker
* Myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within 6 months of the screening period
* Has hemodynamically significant valvular heart disease
* Pregnant, nursing, or planning to be pregnant
* Any serious medical condition that may adversely affect the safety of the participant or the study
* Currently enrolled in another investigational drug or device trial

  2.Angiographic Exclusion Criteria
* Renal artery stenosis (≥50%) or renal artery aneurysm in either renal artery
* History of prior renal artery intervention including balloon angioplasty or stenting
* Multiple renal arteries where the main renal artery is estimated to supply <75% of the kidney
* Main renal arteries with <3 mm diameter or with <20 mm treatable length (by visual estimation)
* Renal artery abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in average 24-hour ambulatory systolic blood pressue at 3 months follow-up | 3 months

SECONDARY OUTCOMES:
Reduction in average 24-hour ambulatory systolic blood pressue at 6 months | 6 months
Change in office systolic blood pressure | 1 month,3 months,6 months and 12 months
Device or procedure related acute adverse events | 1 month,3 months,6 months and 12 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang X, Mahfoud F, Li W, Dong H, Yu J, Yu S, Chen X, Wang P, Li Z, Lauder L, Wang Z, Ji Z, Dong Y, Han B, Zhu Z, Chen Y, Xu J, Zhao X, Fan W, Xie W, Hubbard B, Hu X, Kario K, Gao R. Efficacy and Safety of Catheter-Based Radiofrequency Renal Denervation in Chinese Patients With Uncontrolled Hypertension: The Randomized, Sham-Controlled, Multi-Center Iberis-HTN Trial. Circulation. 2024 Nov 12;150(20):1588-1598. doi: 10.1161/CIRCULATIONAHA.124.069215. Epub 2024 Sep 4. PMID 39229700